CLINICAL TRIAL: NCT03556384
Title: An Open-Label, Phase 2 Efficacy Study of Temozolomide (TMZ) in Advanced Succinate Dehydrogenase (SDH)-Mutant/Deficient Gastrointestinal Stromal Tumor (GIST)
Brief Title: Temozolomide (TMZ) in Advanced Succinate Dehydrogenase (SDH)-Mutant/Deficient Gastrointestinal Stromal Tumor (GIST)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adam Burgoyne, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Adam Burgoyne, MD, PhD, Associate Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180114; FD-R-6334 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Gastrointestinal Stromal Tumors; Sdh; GIST; Cancer
Keywords: cancer; Temozolomide; GIST; SDH-Mutant/Deficient; SDH; Succinate Dehydrogenase
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Hematoma, Subdural; Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TMZ 85 mg/m2 mg orally (Experimental): TMZ 85 mg/m2 mg orally once for 21 days followed by 7 days without treatment in 28 day cycles.
  Treatment will continue for 6 months (with option to continue if benefiting treatment) or until disease progression or unacceptable toxicity (whichever occurs first). All patients will have regular evaluations for assessment of safety parameters. Temozolomide dose may be held and/or modified for the management of adverse treatment effects according to pre-specified criteria. Patients will have radiographic imaging (CT or MRI) every 8 weeks to assess tumor resection.
  An end of treatment visit for clinical evaluations and safety assessments will be performed approximately 28 days after the last dose of study drug. Patients discontinuing study treatment will be followed every 3-6 months for disease recurrence and survival.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Temozolomide 85 mg/m2 will be administered orally for 21 days followed by 7 days without treatment in 28 day cycles.
  Treatment will continue for 6 months (with option to continue if benefiting treatment) or until disease progression or unacceptable toxicity (whichever occurs first). All patients will have regular evaluations for assessment of safety parameters
  Other Names: TEMODAR®

SUMMARY:
Funding Source - FDA OOPD

FDA-approved products for patients with unresectable or metastatic GIST include therapies such as imatinib and sunitinib. Although there are FDA-approved products for the treatment of advanced/metastatic GIST, these therapies are known to be ineffective in the SDH-mutant/deficient subtype and no known effective therapies exist.

The purpose of this study is to investigate SDH-Mutant/Deficient Gastrointestinal Stromal cancer's response to the drug Temozolomide (TMZ) and aim to improve patient outcomes.

Temozolomide is approved by the FDA for the treatment of newly diagnosed glioblastoma multiforme (GBM) and refractory anaplastic astrocytoma cancers.

Temozolomide is considered experimental because it is not approved by the FDA for the treatment of SDH-Mutant/Deficient Gastrointestinal Stromal Tumor.

DETAILED DESCRIPTION:
This oncology study will be a phase 2 study for patients with advanced or metastatic GIST. This study will determine overall response rate at 6 months for TMZ therapy in patients with SDH-mutant/deficient GIST.

Treatment will continue for 6 months (with option to continue if benefiting treatment) or until disease progression or unacceptable toxicity (whichever occurs first). All patients will have regular evaluations for assessment of safety parameters. Temozolomide dose may be held and/or modified for the management of adverse treatment effects according to pre-specified criteria. Patients will have radiographic imaging (CT or MRI) every 8 weeks to assess tumor resection.

An end of treatment visit for clinical evaluations and safety assessments will be performed approximately 28 days (7 days) after the last dose of study drug. Patients discontinuing study treatment will be followed every 3-6 months for disease recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has pathologically confirmed SDH-mutant/deficient GIST.
2. Has recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy.
3. Patient has an ECOG Performance Status of 0-2.
4. Patient has adequate hematologic, hepatic and renal function.
5. Female patient of childbearing potential has a negative serum or urine pregnancy within 72 hours prior to receiving the first dose of study medication.
6. Female patient of childbearing potential agrees to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
7. Male patient with a partner of childbearing potential agrees to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
8. Has measurable or evaluable disease as per RECIST v1.1 (Appendix B).
9. Life expectancy of >12 weeks.

Exclusion Criteria:

1. Patients who have had major surgery within 4 weeks of initiation of study medication.
2. Patients who are receiving other concurrent anti-neoplastic therapy (e.g., chemotherapy, targeted therapy, immunotherapy, or radiotherapy) at the start of study treatment.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. Evidence of severe or uncontrolled systemic diseases [e.g., unstable or uncompensated respiratory, cardiac (including life threatening arrhythmias)].
5. Unresolved toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy except alopecia (if applicable) unless agreed that the patient can be entered after discussion with the Medical Monitor.
6. Presence of cardiac impairment class III and IV definitions; OR history of myocardial infarction/active ischemic heart disease within one year of study entry; OR uncontrolled dysrhythmias; OR poorly controlled angina.
7. Pregnant or breast-feeding females.
8. Medical condition such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
9. Any concurrent condition which in the investigator's opinion makes it undesirable for the subject to participate in this trial or which would jeopardize compliance with the protocol.
10. Patients who cannot swallow oral formulations of the agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 6 months
  To determine overall response rate at 6 months for TMZ therapy in patients with SDH-mutant/deficient GIST

SECONDARY OUTCOMES:
Progression-free survival | 4 years
  Progression-free survival
Overall survival | 4 years
  Overall survival
Adverse events related to TMZ | 6 months
  Description, grade [CTCAE v4.03], and seriousness

CONTACTS AND LOCATIONS:
Overall Officials: Adam Burgoyne, MD, PhD, Principal Investigator — University of California, San Diego; Jason Sicklick, MD, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Miami, Miami, Florida
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No